CLINICAL TRIAL: NCT00917696
Title: A Randomized, Double Blind, Placebo Controlled, Crossover Clinical Trial to Evaluate the Effects of ATP-Induced Pain (AIP) and ATP-induced Dermal Vasodilation (AIDV) by Iontophoresis in Healthy Subjects
Brief Title: Study to Evaluate ATP-induced Pain and ATP-induced Dermal Vasodilation by Iontophoresis (0000-118)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0000-118; 2009_600
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Osteoarthritis Pain
MeSH Terms: interventions — Adenosine Triphosphate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): ATP
  Interventions: Procedure: Comparator: Iontophoresis and Laser Doppler with ATP
- 2 (Placebo Comparator): Saline
  Interventions: Procedure: Comparator: Iontophoresis and Laser Doppler with Saline

INTERVENTIONS:
Procedure: Comparator: Iontophoresis and Laser Doppler with ATP — Iontophoresis treatments with 10 mM ATP (adenosine triphosphate) solution and a current of 0.8 or 1.2 mA. Iontophoresis treatments will last 4 minutes. Laser doppler will be used during the iontophoresis treatments to measure dermal blood flow.
  Arms: 1
Procedure: Comparator: Iontophoresis and Laser Doppler with Saline — Iontophoresis treatments with 20 mM saline solution and a current of 0.8 or 1.2 mA. Iontophoresis treatments will last 4 minutes. Laser doppler will be used during the iontophoresis treatments to measure dermal blood flow.
  Arms: 2

SUMMARY:
This study will evaluate ATP-induced Pain (AIP) and ATP-induced dermal vasodilation (AIDV) as target engagement tools for future development of analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in generally good health
* Subject is willing to abstain from smoking within 24 hours of each iontophoresis treatment and limit smoking to 5 or less cigarettes per week during the study

Exclusion Criteria:

* Subject has a history of dermatitis, psoriasis, or eczema
* Subject has active asthma and/or hay fever at the time of the screening visit
* Subject is unable to refrain from use of analgesics within 3 days prior to each treatment period

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Degree of pain induced by ATP vs. saline iontophoresis | 4 minutes
Increase in blood flow induced by ATP iontophoresis | 8 minutes

SECONDARY OUTCOMES:
Test-retest reproducibility and intra-subject variability of AIP and AIDV | 8 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC